CLINICAL TRIAL: NCT04275115
Title: Interventional, Open-label, One-sequence Study to Investigate the Effects of Multiple Doses of Foliglurax on the Pharmacokinetics of Cytochrome P450 (CYP450) Substrates Caffeine (CYP1A2), Montelukast (CYP2C8), and Midazolam (CYP3A4) in Healthy Subjects
Brief Title: Effects of Repeated Doses of Foliglurax on Drug Metabolizing Enzymes in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18337A
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — foliglurax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foliglurax (Experimental): Foliglurax, iv midazolam and cocktail of CYP450 probe substrates
  Interventions: Drug: Drug Cocktail; Drug: Foliglurax; Drug: midazolam iv

INTERVENTIONS:
Drug: Drug Cocktail — Single oral dose of the cocktail probe substrates (caffeine 200 mg, montelukast 10 mg, midazolam 4 mg)
Drug: Foliglurax — Foliglurax
Drug: midazolam iv — Single intravenous (iv) dose of midazolam 0.025 mg/kg

SUMMARY:
The purpose of this study is to help determine which types of drugs that may interact with foliglurax

DETAILED DESCRIPTION:
This study is designed to evaluate the PK of caffeine, montelukast and midazolam following multiple doses of foliglurax in healthy subjects. The study is divided into four periods:

* Period 1: investigation of the CYP450 probe substrates (caffeine, montelukast, midazolam) alone followed by a 2-day washout before start of Period 2.
* Period 2: administration of foliglurax for 7 days to reach steady state.
* Period 3: administration of the CYP450 probe substrates in combination with foliglurax followed by a 7-day washout before start of Period 4.
* Period 4: investigation of the effects of foliglurax on the PK of the CYP450 probe substrates following washout of foliglurax.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women with a body mass index (BMI) of ≥ 18.5 and ≤ 30 kg/m2 and a minimum body weight of 60 kg for men and 50 kg for women.
* Women of child-bearing potential will have a confirmed non-pregnant and non-lactating status.

Exclusion Criteria:

* The subject has a regular intake of more than 500 mg of caffeine per day or impossibility to stop intake, on holidays for example, without headaches forcing to take caffeine again.

Other in- and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
AUC0-inf | Day 1 and 11 for midazolam iv and Day 2,12 and 20 for oral cocktail probe substrates
  Area under the plasma concentration-time curve from zero to infinity for midazolam after iv administration and for all oral cocktail probe substrates
Cmax | Day 1 and 11 for midazolam iv and Day 2,12 and 20 for oral cocktail probe substrates
  Maximum observed plasma concentration of midazolam after iv administration and for all oral cocktail probe substrates

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided